CLINICAL TRIAL: NCT04938804
Title: Non-risk Based Lung Cancer Screening With One-time Low-dose Computed Tomography: a Prospective Cohort Study
Brief Title: Non-risk Based Lang Cancer Screening With a One-off LDCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GZLUNG
Record Dates: First submitted 2021-06-12; First posted 2021-06-24 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: Screening
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening group (Experimental)
  Interventions: Device: Low-dose computed tomography

INTERVENTIONS:
Device: Low-dose computed tomography — The Low-dose computed tomography is conducted according to the guideline suggested by American College of Radiology.

SUMMARY:
Guangzhou Lung-Care Project is a single-arm, prospective cohort study using one-time low-dose computed tomography for the early detection of LC, recruiting residents aged 40-74 years from four communities in Guangzhou between 2015 and 2021.The primary outcome was LC detection rate in eligible participants without restrictions based on high-risk factors and the proportion of stage I LC cases, and to investigate the various factors associated with the development of LC.

DETAILED DESCRIPTION:
Guangzhou Lung-Care Project is a single-arm, prospective cohort study using one-time low-dose computed tomography for the early detection of LC, recruiting residents aged 40-74 years from four communities in Guangzhou between 2015 and 2021. Follow-up for post-screening management and survival was recorded. The primary outcome was LC detection rate in eligible participants without restrictions based on high-risk factors and the proportion of stage I LC cases, and to investigate the various factors associated with the development of LC. Additionally, we compared the detection rates of LC and the proportion of stage I LC cases between "high-risk" and "non-high-risk" groups according to the National Comprehensive Cancer Network (NCCN) guidelines and Chinese guideline.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 40 years among the residents in Guangzhou

Exclusion Criteria:

* Persons who had a diagnosis or treatment related to LC within the past 5 years, had undergone chest CT within the past year, or had significant cancer-related symptoms (e.g., hemoptysis, dyspnea, inability to climb two flights of stairs).

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11000 (Estimated)
Dates: Start 2015-12-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The detection rate of lung cancer | 11 years
  Lung cancer detection rate in eligible participants without restrictions based on high-risk factors and the proportion of stage I LC cases.
To investigate the various factors associated with the development of lung cancer | 11 years
  To investigate the various factors associated with the development of lung cancer

SECONDARY OUTCOMES:
Detection rates of lung cancer and the proportion of stage I lung cancer cases between "high-risk" and "non-high-risk" groups | 11 years
  The detection rate of lung cancer among people with "high-risk" and "non-high-risk"factors
Cost-effectiveness ratio (costs of examinations, diagnoses, and treatments) | 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Wenhua Liang, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ye W, Fu W, Li C, Li J, Xiong S, Cheng B, Xu B, Wang Q, Feng Y, Chen P, He J, Liang W. Diameter thresholds for pure ground-glass pulmonary nodules at low-dose CT screening: Chinese experience. Thorax. 2025 Jan 17;80(2):76-85. doi: 10.1136/thorax-2024-221642. PMID 39689940